CLINICAL TRIAL: NCT00364585
Title: A Prospective Evaluation of the GreenLight Model 120 Laser System for the Treatment of Benign Prostatic Hyperplasia
Brief Title: A Prospective Evaluation of the GreenLight Model 120 Laser
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0604008494; 0000022806
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

INTERVENTIONS:
Device: GreenLight Model 120 Laser System

SUMMARY:
The purpose of this study is to evaluate the performance of the GreenLight™ model 120 delivering higher average power to allow for more flexibility in the working distance of the delivery device with the same power density to tissue as that of the current GreenLight model. In addition this study will examine the Laserscope GDD (guided delivery device) that has been designed exclusively for use with the GreenLight™ model 120.

DETAILED DESCRIPTION:
Benign Prostatic Hyperplasia (BPH) refers to a medical condition which occurs in aging men where the prostate gland is enlarged preventing the free flow of urine. This causes symptoms of frequent urination, constant feeling of urgency to go to the bathroom, and difficulty passing urine due to the obstruction caused by the enlarged gland. The incidence (number of new cases) of BPH increases from 40% among males between the ages of 50 and 60 years to 90% among males older than 80 years of age. Treatment of BPH is currently undergoing intense scrutiny due to the cost and morbidity (complications and disability due to the procedure) associated with the "gold standard" treatment, Transurethral Resection of the Prostate (TURP). The TURP procedure has established its place as a standard of care for BPH due to its exceptional clinical efficacy and established long-term durability. Despite the clinical prowess of TURP, there remain significant concerns regarding the relatively high incidence of postoperative morbidity and the significant economic burden on world healthcare systems. Laser vaporization prostatectomy, on the other hand, has developed into a relatively new technological advance that has been utilized with favorable outcomes for more than a decade.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be male and over the age of 40 years.
2. Subjects must present with symptomatic/obstructive symptoms secondary to BPH requiring surgical intervention, diagnosed using standard clinical practices (uroflowmetry).
3. Subjects must present with LUTS secondary to BPH > 3 months in duration.
4. IPPS symptom score value of > 12.
5. Prostate size, as measured by transrectal ultrasonography, between 15 and 300 cc.
6. Subjects that are in retention may be enrolled in the study provided that it is documented the primary cause of the retention is BPH.
7. ASA classification of physical status, class 1-3.
8. Subjects must read, understand, and sign the Informed Consent.
9. Subjects must be willing and able to comply with all follow-up requirements.

Exclusion Criteria:

1. Unstable cardiopulmonary disorder, previously or recently diagnosed by standard methods.
2. Subjects with a recent myocardial infarction or coronary artery stent placement.
3. Subjects with systemic diseases that cause significant neurogenic lower urinary dysfunction.
4. Subjects who have had major pelvic fractures that involved damage to the external urinary sphincter.
5. Subjects who have recently completed definitive radiation therapy for prostate cancer.
6. Subjects with prostate cancer who are considering brachytherapy (radioactive seed implantation) or cryotherapy as part of their definitive treatment.
7. Subjects must not have active localized or systemic infections; including active urinary tract infection.
8. Subjects with confirmed atonic bladders and/or neurogenic bladders, reflex dyssynergia, detrusor hyporeflexia/areflexia.
9. Subjects diagnosed with active urethral strictures, bladder neck contracture, acute prostatitis affecting bladder function.
10. Serum prostate specific antigen level > 4 ng/ml, requiring prostate needle biopsy, and resultant positive pathology for malignancy of the prostate.
11. Subjects with confirmed or suspected malignancy of the prostate or bladder.
12. Subjects with renal ectasia by renal ultrasound.
13. Immunocompromised subjects and deemed unfit for laser vaporization as determined by the attending physician.
14. Any disorder or conditions of the subject that the investigator believes will contraindicate their inclusion in the study.
15. Subjects who refuse to sign the Informed Consent document and/or comply with all follow-up requirements.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-05; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of the GreenLightÔ Model 120 Laser for the treatment (PVP)

SECONDARY OUTCOMES:
To evaluate the effectiveness of the Laserscope GDD

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Te, MD, Principal Investigator — Cornell University
Locations (1):
- New York-Presbyterian Hospital Cornell Univeristy, New York, New York, United States